CLINICAL TRIAL: NCT04618887
Title: A Comparative Study of GPI's DBS and Pallidotomy in the Treatment of Meige Syndrome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Ruen, PekingUPH, Peking University People's Hospital
Other Study IDs: MeigeSyndrome
Record Dates: First submitted 2020-11-01; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Meige Syndrome; Meigs Syndrome; Meige Disease; Meig Syndrome; Blepharospasm; Blepharospasm of Left Eyelid; Blepharospasm of Right Eyelid; Blepharospasm of Both Eyelids; Blepharospasm Oromandibular Dystonia
Keywords: deep brain stimulation; DBS; DBNL; GPi; pallidotomy
MeSH Terms: conditions — Meige Syndrome; Meigs Syndrome; Lymphedema, Hereditary, II; Blepharospasm | interventions — Pallidotomy; Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Meige sydrome patients
  Interventions: Procedure: pallidotomy; Procedure: deep brain stimulation

INTERVENTIONS:
Procedure: pallidotomy — deep brain nuclei lesion of GPi
Procedure: deep brain stimulation — deep brain stimulation of GPi

SUMMARY:
In this study, we will compare the degree of postoperative symptom improvement, postoperative complication rate, postoperative quality of life improvement degree of patients with Meige syndrome undergoing pallidotomy (unilateral globus palliotomy) and deep brain stimulation (unilateral globus pallidus) ,in order to get the conclusion of the comparison of the clinical efficacy of the two surgical plans. In addition, possible predictive factors such as age, gender, age of onset, length of disease course, scale baseline score, preoperative brain PET-CT function analysis and other possible predictive factors are added for analysis, in order to find predictive factors that can guide the choice of surgical options.

ELIGIBILITY:
Inclusion Criteria:

* Patients confirmed Meige sydrome

Exclusion Criteria:

* Patients who cannot finish the neurosurgery or the postoperative evaluation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lack of incidence of Meige sydrome，and also lack of efficient of DBS or pallidotomy of Meige Syndrome. We try to collect more data as we can. We initially established a population of 100.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Symptom | 2 years
  spasm of eyelid
complications | 2 years
  Postoperative complications

SECONDARY OUTCOMES:
quality of life | 2 years
  Evaluate using SF-36
depression scale | 2 years
  Evaluate using Hamilton Depression Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided